CLINICAL TRIAL: NCT04663802
Title: Implementation of Nudges to Promote Utilization of Low Tidal Volume Ventilation (INPUT) Study
Acronym: INPUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 833400; 1R01HL141608-01A1 (NIH)
Record Dates: First submitted 2020-06-05; First posted 2020-12-11 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: ARDS; Critical Illness; Acute Respiratory Distress Syndrome; Acute Respiratory Failure
Keywords: mechanical ventilation; lung-protective ventilation
MeSH Terms: conditions — Critical Illness; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Usual care (No Intervention): This arm will have no interventions and standard of care practices will be in place.
- Default order set (Active Comparator): This arm will have the default order set implementation strategy
  Interventions: Behavioral: Default order set
- Physician-targeted accountable justification (Active Comparator): This arm will have the physician-targeted accountable justification implementation strategy
  Interventions: Behavioral: Physician-targeted accountable justification
- Default order set + RT-targeted accountable justification (Active Comparator): This arm will have the default order set and respiratory therapist-targeted accountable justification
  Interventions: Behavioral: Default order set; Behavioral: Respiratory therapist (RT)-targeted accountable justification
- Physician-targeted accountable justification + RT-targeted accountable justification (Active Comparator): This arm will have the default order set and respiratory therapist-targeted accountable justification
  Interventions: Behavioral: Physician-targeted accountable justification; Behavioral: Respiratory therapist (RT)-targeted accountable justification

INTERVENTIONS:
Behavioral: Default order set — With the default order set strategy, some mechanical ventilation order settings will be pre-populated to be consistent with LPV, including the mode and tidal volume, automatically calculated as 6 milliliters per kilogram of predicted body weight (cc/kg PBW; as determined by each patient's height and gender). The physician will have the option to opt out of any of the specified LPV settings and select other values.
  Arms: Default order set; Default order set + RT-targeted accountable justification
Behavioral: Physician-targeted accountable justification — When a physician enters a mechanical ventilation order for a tidal volume that is greater than 6 cc/kg PBW, an alert will appear requiring the physician to enter a reason for choosing a setting inconsistent with LPV. Clinicians will be instructed to provide a reason for deviation from LPV settings and that their response will be maintained in the medical record. The physician will not be able to sign the mechanical ventilation order set until after a response is entered.
  Arms: Physician-targeted accountable justification; Physician-targeted accountable justification + RT-targeted accountable justification
Behavioral: Respiratory therapist (RT)-targeted accountable justification — If an RT enters a tidal volume in a flowsheet documentation field value greater than 6 cc/kg PBW, an alert will appear requiring them to enter a reason for entering a setting inconsistent with LPV. Clinicians will be instructed to provide a reason for deviation from LPV settings and that their response will be maintained in the medical record. The RT will not be able to save the documentation in the EHR until after a response is entered.
  Arms: Default order set + RT-targeted accountable justification; Physician-targeted accountable justification + RT-targeted accountable justification

SUMMARY:
This study is a large pragmatic stepped-wedge trial of electronic health record (EHR)-based implementation strategies informed by behavioral economic principles to increase lung-protective ventilation (LPV) utilization among all mechanically ventilated (MV), adult patients. The study will compare the standard approach to managing MV across 12 study Intensive Care Units (ICUs) within University of Pennsylvania Health System (UPHS) versus interventions prompting physicians and respiratory therapists (RTs) to employ LPV settings promote LPV utilization among all MV patients.

DETAILED DESCRIPTION:
The study is a 5-arm, stepped-wedge cluster randomized trial of electronic health record (EHR)-based implementation strategies set in 12 community and academic intensive care units (ICUs) in 5 hospitals of UPHS all currently using an EHR-based algorithm to identify patients with Acute Respiratory Distress Syndrome (ARDS) and prompt physicians to employ LPV will sequentially add two of three EHR-based implementation strategies to further promote LPV utilization among all MV patients. ICUs will be randomly assigned to first receive either a default order set (Strategy A) or physician-targeted accountable justification strategy (Strategy B). ICUs will be assigned to one of six wedges using computerized random-number generation, thereby determining the date on which they adopt their assigned EHR-based strategy. The first wedge will begin in the fourth month of the trial phase, so that all hospitals will contribute a minimum of 3 months of data prior to having adopted the implementation strategy. Six months after adoption, ICUs will add on an accountable justification strategy targeting respiratory therapists (RT; Strategy C). By the end of the 27-month study period, all hospitals will have been utilizing two strategies in combination for at least 3 months. This design enables comparisons of outcomes before and after implementation within ICUs, as well as at a given point in time among ICUs which will have been randomly assigned to different strategies. During the two months after the implementation strategy rolls out in each ICU, researchers will perform semi-structured interviews of all physicians and RTs who staff study ICUs. After intervention period, there will be a 6-month observational period where trial monitoring will cease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and over; AND
2. Admission to 1 of the 12 participating ICUs; AND
3. Undergoing mechanical ventilation

Exclusion Criteria:

1. The episode of MV lasts less than 12 hours, because we believe that the evidence-based practice may not apply to these patients nor alter their outcomes.
2. The patient is on minimal settings for the entirety of MV, defined as a spontaneous mode (e.g., pressure support ventilation) with pressure support <10 Centimeters of Water Column (cmH2O), AND positive end-expiratory pressure (PEEP) <8 cmH20, AND fraction of inspired oxygen (FiO2) <50%, because the clinical significance of spontaneous tidal volumes is unknown and low tidal volumes may not be beneficial or desirable.
3. Goals of care are documented as comfort measures only (as identified through their "code status" field in the EHR) during the first 72 hours during episode of MV, because mechanical ventilation is managed differently during care focused exclusively on comfort and low tidal volume ventilation may not be appropriate, nor would it likely influence clinical outcomes.
4. There is no height documented in the EHR at the time of initiation of MV, because we will be unable to estimate ideal body weight, a necessary parameter to calculate the primary outcome, and because they will not receive the interventions.
5. The height documented is less than 4 feet, because the formula for ideal body weight does not hold true below this height.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7342 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meeta Kerlin, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (5):
- United States (5):
  - Princeton Medical Center, Plainsboro, New Jersey
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie published results will be made available to other researchers, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 9 months after publication and up to 36 months following publication. After 36 months the data will be available in our University's data warehouse but without support, except for deposited metadata.
Access Criteria: Proposals for data use will be reviewed by Principal Investigator and independent review boards (such as Institutional Review Board and Data Safety and Monitoring Board). Approved data requestors will need to sign data use agreements to access and use data
URL: https://www.pair.upenn.edu

REFERENCES:
- [Derived] Kerlin MP, Small D, Fuchs BD, Mikkelsen ME, Wang W, Tran T, Scott S, Belk A, Silvestri JA, Klaiman T, Halpern SD, Beidas RS. Implementing nudges to promote utilization of low tidal volume ventilation (INPUT): a stepped-wedge, hybrid type III trial of strategies to improve evidence-based mechanical ventilation management. Implement Sci. 2021 Aug 10;16(1):78. doi: 10.1186/s13012-021-01147-7. PMID 34376233

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Intensive care units (ICUs)
Groups:
- Strategy A+C, Wedge 1 (ICU #1): 3 months of usual care followed by 6 months with Strategy A alone (a nudge embedded in the order panel including pre-specified settings for mechanical ventilation including tidal volume of 6 milliliters per kilogram predicted body weight [cc/kg PBW]that can be opted out of by the ordering clinician at any time with a click), followed by 18 months with Strategy A+C (strategy A as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy B+C, Wedge 1 (ICU #2): 3 months of usual care followed by 6 months with Strategy B alone (a nudge embedded in the order panel requiring a free-text justification if a tidal volume greater than 6.5 cc/kg PBW is ordered), followed by 18 months with Strategy B+C (strategy B as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy A+C, Wedge 2 (ICU #3): 6 months of usual care followed by 6 months with Strategy A alone (a nudge embedded in the order panel including pre-specified settings for mechanical ventilation including tidal volume of 6 cc/kg PBW that can be opted out of by the ordering clinician at any time with a click), followed by 15 months with Strategy A+C (strategy A as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy B+C, Wedge 2 (ICU #4): 6 months of usual care followed by 6 months with Strategy B alone (a nudge embedded in the order panel requiring a free-text justification if a tidal volume greater than 6.5 cc/kg PBW is ordered), followed by 15 months with Strategy B+C (strategy B as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg PBW into the flowsheet).
- Strategy A+C, Wedge 3 (ICU #5): 9 months of usual care followed by 6 months with Strategy A alone (a nudge embedded in the order panel including pre-specified settings for mechanical ventilation including tidal volume of 6 cc/kg PBW that can be opted out of by the ordering clinician at any time with a click), followed by 12 months with Strategy A+C (strategy A as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy B+C, Wedge 3 (ICU #6): 9 months of usual care followed by 6 months with Strategy B alone (a nudge embedded in the order panel requiring a free-text justification if a tidal volume greater than 6.5 cc/kg PBW is ordered), followed by 12 months with Strategy B+C (strategy B as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy A+C, Wedge 4 (ICU #7): 12 months of usual care followed by 6 months with Strategy A alone (a nudge embedded in the order panel including pre-specified settings for mechanical ventilation including tidal volume of 6 cc/kg PBW that can be opted out of by the ordering clinician at any time with a click), followed by 9 months with Strategy A+C (strategy A as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy B+C, Wedge 4 (ICU #8): 12 months of usual care followed by 6 months with Strategy B alone (a nudge embedded in the order panel requiring a free-text justification if a tidal volume greater than 6.5 cc/kg PBW is ordered), followed by 9 months with Strategy B+C (strategy B as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy A+C, Wedge 5 (ICU #9): 15 months of usual care followed by 6 months with Strategy A alone (a nudge embedded in the order panel including pre-specified settings for mechanical ventilation including tidal volume of 6 cc/kg PBW that can be opted out of by the ordering clinician at any time with a click), followed by 6 months with Strategy A+C (strategy A as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy B+C, Wedge 5 (ICU #10): 15 months of usual care followed by 6 months with Strategy B alone (a nudge embedded in the order panel requiring a free-text justification if a tidal volume greater than 6.5 cc/kg PBW is ordered), followed by 6 months with Strategy B+C (strategy B as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy A+C, Wedge 6 (ICU #11): 18 months of usual care followed by 6 months with Strategy A alone (a nudge embedded in the order panel including pre-specified settings for mechanical ventilation including tidal volume of 6 cc/kg PBW that can be opted out of by the ordering clinician at any time with a click), followed by 3 months with Strategy A+C (strategy A as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
- Strategy B+C, Wedge 6 (ICU #12): 18 months of usual care followed by 6 months with Strategy B alone (a nudge embedded in the order panel requiring a free-text justification if a tidal volume greater than 6.5 cc/kg PBW is ordered), followed by 3 months with Strategy B+C (strategy B as above combined with nudge that requires that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6.5 cc/kg PBW into the flowsheet).
Period: Step 1: 2/22/2021 to 5/16/2021
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 85; 1 Intensive care units (ICUs) | 91; 1 Intensive care units (ICUs) | 30; 1 Intensive care units (ICUs) | 28; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 53; 1 Intensive care units (ICUs) | 104; 1 Intensive care units (ICUs) | 66; 1 Intensive care units (ICUs) | 141; 1 Intensive care units (ICUs) | 55; 1 Intensive care units (ICUs) | 58; 1 Intensive care units (ICUs) | 40; 1 Intensive care units (ICUs)
Completed | 85; 1 Intensive care units (ICUs) | 91; 1 Intensive care units (ICUs) | 30; 1 Intensive care units (ICUs) | 28; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 53; 1 Intensive care units (ICUs) | 104; 1 Intensive care units (ICUs) | 66; 1 Intensive care units (ICUs) | 141; 1 Intensive care units (ICUs) | 55; 1 Intensive care units (ICUs) | 58; 1 Intensive care units (ICUs) | 40; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 2: 5/17/2021 to 8/15/2021
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 64; 1 Intensive care units (ICUs) | 99; 1 Intensive care units (ICUs) | 39; 1 Intensive care units (ICUs) | 24; 1 Intensive care units (ICUs) | 64; 1 Intensive care units (ICUs) | 40; 1 Intensive care units (ICUs) | 95; 1 Intensive care units (ICUs) | 61; 1 Intensive care units (ICUs) | 132; 1 Intensive care units (ICUs) | 46; 1 Intensive care units (ICUs) | 62; 1 Intensive care units (ICUs) | 40; 1 Intensive care units (ICUs)
Completed | 64; 1 Intensive care units (ICUs) | 99; 1 Intensive care units (ICUs) | 39; 1 Intensive care units (ICUs) | 24; 1 Intensive care units (ICUs) | 64; 1 Intensive care units (ICUs) | 40; 1 Intensive care units (ICUs) | 95; 1 Intensive care units (ICUs) | 61; 1 Intensive care units (ICUs) | 132; 1 Intensive care units (ICUs) | 46; 1 Intensive care units (ICUs) | 62; 1 Intensive care units (ICUs) | 40; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 3: 8/16/2021 to 11/14/2021
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 88; 1 Intensive care units (ICUs) | 76; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 21; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 91; 1 Intensive care units (ICUs) | 66; 1 Intensive care units (ICUs) | 124; 1 Intensive care units (ICUs) | 52; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 53; 1 Intensive care units (ICUs)
Completed | 88; 1 Intensive care units (ICUs) | 76; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 21; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 91; 1 Intensive care units (ICUs) | 66; 1 Intensive care units (ICUs) | 124; 1 Intensive care units (ICUs) | 52; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 53; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 4: 11/15/2021 to 2/20/2022
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 76; 1 Intensive care units (ICUs) | 86; 1 Intensive care units (ICUs) | 56; 1 Intensive care units (ICUs) | 49; 1 Intensive care units (ICUs) | 71; 1 Intensive care units (ICUs) | 47; 1 Intensive care units (ICUs) | 97; 1 Intensive care units (ICUs) | 68; 1 Intensive care units (ICUs) | 151; 1 Intensive care units (ICUs) | 69; 1 Intensive care units (ICUs) | 83; 1 Intensive care units (ICUs) | 82; 1 Intensive care units (ICUs)
Completed | 76; 1 Intensive care units (ICUs) | 86; 1 Intensive care units (ICUs) | 56; 1 Intensive care units (ICUs) | 49; 1 Intensive care units (ICUs) | 71; 1 Intensive care units (ICUs) | 47; 1 Intensive care units (ICUs) | 97; 1 Intensive care units (ICUs) | 68; 1 Intensive care units (ICUs) | 151; 1 Intensive care units (ICUs) | 69; 1 Intensive care units (ICUs) | 83; 1 Intensive care units (ICUs) | 82; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 5: 2/21/2022 to 5/15/2022
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 71; 1 Intensive care units (ICUs) | 71; 1 Intensive care units (ICUs) | 41; 1 Intensive care units (ICUs) | 32; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 27; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 58; 1 Intensive care units (ICUs) | 132; 1 Intensive care units (ICUs) | 48; 1 Intensive care units (ICUs) | 70; 1 Intensive care units (ICUs) | 51; 1 Intensive care units (ICUs)
Completed | 71; 1 Intensive care units (ICUs) | 71; 1 Intensive care units (ICUs) | 41; 1 Intensive care units (ICUs) | 32; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 27; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 58; 1 Intensive care units (ICUs) | 132; 1 Intensive care units (ICUs) | 48; 1 Intensive care units (ICUs) | 70; 1 Intensive care units (ICUs) | 51; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 6: 5/16/2022 to 8/21/2022
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 66; 1 Intensive care units (ICUs) | 74; 1 Intensive care units (ICUs) | 39; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 71; 1 Intensive care units (ICUs) | 36; 1 Intensive care units (ICUs) | 76; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 128; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 63; 1 Intensive care units (ICUs) | 59; 1 Intensive care units (ICUs)
Completed | 66; 1 Intensive care units (ICUs) | 74; 1 Intensive care units (ICUs) | 39; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 71; 1 Intensive care units (ICUs) | 36; 1 Intensive care units (ICUs) | 76; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 128; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 63; 1 Intensive care units (ICUs) | 59; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 7: 8/22/2022 to11/20/2022
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 78; 1 Intensive care units (ICUs) | 75; 1 Intensive care units (ICUs) | 51; 1 Intensive care units (ICUs) | 48; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 37; 1 Intensive care units (ICUs) | 86; 1 Intensive care units (ICUs) | 78; 1 Intensive care units (ICUs) | 159; 1 Intensive care units (ICUs) | 70; 1 Intensive care units (ICUs) | 77; 1 Intensive care units (ICUs) | 64; 1 Intensive care units (ICUs)
Completed | 78; 1 Intensive care units (ICUs) | 75; 1 Intensive care units (ICUs) | 51; 1 Intensive care units (ICUs) | 48; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 37; 1 Intensive care units (ICUs) | 86; 1 Intensive care units (ICUs) | 78; 1 Intensive care units (ICUs) | 159; 1 Intensive care units (ICUs) | 70; 1 Intensive care units (ICUs) | 77; 1 Intensive care units (ICUs) | 64; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 8: 11/21/2022 to 2/19/2023
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 71; 1 Intensive care units (ICUs) | 88; 1 Intensive care units (ICUs) | 41; 1 Intensive care units (ICUs) | 46; 1 Intensive care units (ICUs) | 80; 1 Intensive care units (ICUs) | 48; 1 Intensive care units (ICUs) | 103; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 117; 1 Intensive care units (ICUs) | 80; 1 Intensive care units (ICUs) | 55; 1 Intensive care units (ICUs) | 86; 1 Intensive care units (ICUs)
Completed | 71; 1 Intensive care units (ICUs) | 88; 1 Intensive care units (ICUs) | 41; 1 Intensive care units (ICUs) | 46; 1 Intensive care units (ICUs) | 80; 1 Intensive care units (ICUs) | 48; 1 Intensive care units (ICUs) | 103; 1 Intensive care units (ICUs) | 67; 1 Intensive care units (ICUs) | 117; 1 Intensive care units (ICUs) | 80; 1 Intensive care units (ICUs) | 55; 1 Intensive care units (ICUs) | 86; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)
Period: Step 9: 2/20/2023 to 5/15/2023
Arm/Group | Strategy A+C, Wedge 1 (ICU #1) | Strategy B+C, Wedge 1 (ICU #2) | Strategy A+C, Wedge 2 (ICU #3) | Strategy B+C, Wedge 2 (ICU #4) | Strategy A+C, Wedge 3 (ICU #5) | Strategy B+C, Wedge 3 (ICU #6) | Strategy A+C, Wedge 4 (ICU #7) | Strategy B+C, Wedge 4 (ICU #8) | Strategy A+C, Wedge 5 (ICU #9) | Strategy B+C, Wedge 5 (ICU #10) | Strategy A+C, Wedge 6 (ICU #11) | Strategy B+C, Wedge 6 (ICU #12)
Started | 72; 1 Intensive care units (ICUs) | 65; 1 Intensive care units (ICUs) | 35; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 43; 1 Intensive care units (ICUs) | 85; 1 Intensive care units (ICUs) | 56; 1 Intensive care units (ICUs) | 103; 1 Intensive care units (ICUs) | 55; 1 Intensive care units (ICUs) | 53; 1 Intensive care units (ICUs) | 43; 1 Intensive care units (ICUs)
Completed | 72; 1 Intensive care units (ICUs) | 65; 1 Intensive care units (ICUs) | 35; 1 Intensive care units (ICUs) | 38; 1 Intensive care units (ICUs) | 73; 1 Intensive care units (ICUs) | 43; 1 Intensive care units (ICUs) | 85; 1 Intensive care units (ICUs) | 56; 1 Intensive care units (ICUs) | 103; 1 Intensive care units (ICUs) | 55; 1 Intensive care units (ICUs) | 53; 1 Intensive care units (ICUs) | 43; 1 Intensive care units (ICUs)
Not Completed | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs) | 0; 0 Intensive care units (ICUs)

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care (Baseline): This arm will have no interventions and standard of care practices will be in place.
  Standard of Care: ICUs and clinicians will deliver standard of care to patients with no intervention
- Default Order Set: This arm will have the default order set implementation strategy
  Default order set: With the default order set strategy, some mechanical ventilation order settings will be pre-populated to be consistent with LPV, including the mode and tidal volume, automatically calculated as 6 cc/kg of the patient's ideal body weight (as determined by each patient's height and gender, which are entered into the EHR on admission). The physician will have the option to opt out of any of the specified LPV settings and select other values.
- Physician-targeted Accountable Justification: This arm will have the physician-targeted accountable justification implementation strategy
  Physician-targeted accountable justification: When a physician enters a mechanical ventilation order for a tidal volume that is greater than 6 cc/kg ideal body weight, an alert will appear requiring the physician to enter a reason for choosing a setting inconsistent with LPV. Clinicians will be instructed to provide a reason for deviation from LPV settings and that their response will be maintained in the medical record. The physician will not be able to sign the mechanical ventilation order set until after a response is entered.
- Default Order Set + RT-targeted Accountable Justification: This arm will have the default order set and physician-targeted accountable justification
  Default order set: With the default order set strategy, some mechanical ventilation order settings will be pre-populated to be consistent with LPV, including the mode and tidal volume, automatically calculated as 6 cc/kg of the patient's ideal body weight (as determined by each patient's height and gender, which are entered into the EHR on admission). The physician will have the option to opt out of any of the specified LPV settings and select other values.
  RT-targeted accountable justification: This strategy will require that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg into the flowsheet, similar to the physician-targeted accountable justification strategy.
- Physician-targeted Accountable Justification + RT-targeted Accountable Justification: This arm will have both the physician-targeted and respiratory therapist-targeted accountable justification interventions
  Physician-targeted accountable justification: When a physician enters a mechanical ventilation order for a tidal volume that is greater than 6 cc/kg ideal body weight, an alert will appear requiring the physician to enter a reason for choosing a setting inconsistent with LPV. Clinicians will be instructed to provide a reason for deviation from LPV settings and that their response will be maintained in the medical record. The physician will not be able to sign the mechanical ventilation order set until after a response is entered.
  RT-targeted accountable justification: This strategy will require that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg into the flowsheet, similar to the physician-targeted accountable justification strategy.
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Baseline) | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification | Total
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196 | 7342
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [50 to 71] | 61 [48 to 71] | 64 [54 to 74] | 63 [51 to 71] | 63 [53 to 72] | 63 [51 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1199 | 336 | 325 | 569 | 512 | 2941
  Male | 1777 | 620 | 409 | 911 | 684 | 4401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 13 | 11 | 6 | 2 | 57
  Not Hispanic or Latino | 2853 | 915 | 710 | 1452 | 1186 | 7116
  Unknown or Not Reported | 98 | 28 | 13 | 22 | 8 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 2 | 3 | 1 | 15
  Asian | 96 | 32 | 43 | 37 | 60 | 268
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 4 | 4 | 2 | 11
  Black or African American | 1063 | 328 | 250 | 521 | 407 | 2569
  White | 1496 | 455 | 381 | 671 | 607 | 3610
  More than one race | 11 | 5 | 3 | 3 | 4 | 26
  Unknown or Not Reported | 304 | 132 | 51 | 241 | 115 | 843
Region of Enrollment [Number; unit: participants]
  United States | 2976 | 956 | 734 | 1480 | 1196 | 7342

OUTCOME MEASURES:

1. Primary Outcome: Fidelity to LPV
Description: percentage of time that a patient is exposed to tidal volume <6.5 cc/kg ideal body weight
Time Frame: up to 72 hours, from initiation of mechanical ventilation in a study ICU until discontinuation of mechanical ventilation
Measure: Median (Inter-Quartile Range); unit: Percentage of time during first 72 hours
Groups:
- Standard of Care: This arm will have no interventions and standard of care practices will be in place.
  Standard of Care: ICUs and clinicians will deliver standard of care to patients with no intervention
- Physician-targeted Accountable Justification + RT-targeted Accountable Justification: This arm will have the default order set and respiratory therapist-targeted accountable justification
  RT-targeted accountable justification: This strategy will require that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg into the flowsheet, similar to the physician-targeted accountable justification strategy.
  physician-targeted accountable justification: When a physician enters a mechanical ventilation order for a tidal volume that is greater than 6 cc/kg ideal body weight, an alert will appear requiring the physician to enter a reason for choosing a setting inconsistent with LPV. Clinicians will be instructed to provide a reason for deviation from LPV settings and that their response will be maintained in the medical record. The physician will not be able to sign the mechanical ventilation order set until after a response is entered.
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
Percentage of time during first 72 hours | 43.3 [0 to 100] | 19.1 [0 to 98.3] | 83.9 [0.5 to 100] | 31.0 [0 to 99.5] | 67.8 [0 to 100]

2. Secondary Outcome: Total Duration of Exposure to Tidal Volume >8 cc/kg PBW
Description: Total duration of exposure to tidal volume greater than 8 cc/kg PBW, in hours. The time frame for follow-up is based on the total duration of IMV during the total follow-up period of 30 days. Note it is intentionally different from the time frame of the primary outcome variable, which focuses on the initial 72 hours, as the period most likely to be influenced by the study interventions.
Time Frame: from initiation to discontinuation of mechanical ventilation in the study ICU, up to 720 hours (30 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
hours | 0.08 [0 to 10.47] | 0.51 [0 to 10.81] | 0 [0 to 6.45] | 0.37 [0 to 11.06] | 0.09 [0 to 7.98]

3. Secondary Outcome: Total Duration of Exposure to Tidal Volume >10 cc/kg PBW
Description: Total duration of exposure to tidal volume greater than 10 cc/kg PBW, in hours. The time frame for follow-up is based on the total duration of IMV during the total follow-up period of 30 days. Note it is intentionally different from the time frame of the primary outcome variable, which focuses on the initial 72 hours, as the period most likely to be influenced by the study interventions.
Time Frame: from initiation to discontinuation of mechanical ventilation in the study ICU, up to 720 hours (30 days)
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Default Order Set + RT-targeted Accountable Justification: Default order set: With the default order set strategy, some mechanical ventilation order settings will be pre-populated to be consistent with LPV, including the mode and tidal volume, automatically calculated as 6 cc/kg of the patient's ideal body weight (as determined by each patient's height and gender, which are entered into the EHR on admission). The physician will have the option to opt out of any of the specified LPV settings and select other values.
  RT-targeted accountable justification: This strategy will require that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg into the flowsheet, similar to the physician-targeted accountable justification strategy.
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
hours | 0 [0 to 1] | 0 [0 to 1.54] | 0 [0 to 0.25] | 0 [0 to 1.32] | 0 [0 to 1.06]

4. Secondary Outcome: Initial Tidal Volume Administered
Description: Binary variable for whether initial tidal volume (first documented value after initiation of mechanical ventilation in a study ICU) is less than or equal to 6.5 milliliters per kilogram of predicted body weight (cc/kg PBW)
Time Frame: within 24 hours of initiation of mechanical ventilation in a study ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
Participants
  > 6.5 cc/kg PBW | 1628 | 539 | 347 | 822 | 562
  < or equal to 6.5 cc/kg PBW | 1348 | 417 | 387 | 658 | 634

5. Secondary Outcome: Initial Plateau Pressure (Pplat)>30 Centimeters of Water (cm H2O)
Description: Binary variable for whether initial plateau pressure (Pplat) > 30 cm H2O (first documented value after initiation of mechanical ventilation in a study ICU)
Time Frame: within 24 hours of initiation of mechanical ventilation in a study ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
Participants
  >30 | 126 | 26 | 37 | 34 | 43
  < 30 | 2310 | 806 | 507 | 1187 | 903
  missing | 540 | 124 | 190 | 259 | 250

6. Secondary Outcome: Hospital Mortality
Description: All-cause mortality occurring during hospitalization.
Time Frame: All-cause mortality as a study outcome was assessed through hospital discharge, up to 720 hours (30 days); all adverse events (including mortality) were assessed though 24 hours after initiation of mechanical ventilation.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
Participants | 977 | 294 | 268 | 417 | 437

7. Secondary Outcome: ICU-free Days
Description: days alive and not admitted to an ICU; composite of ICU length of stay and death
Time Frame: from time of first eligibility to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
days | 18 [0 to 26] | 16 [0 to 25] | 18.5 [0 to 26] | 19 [0 to 26] | 18 [0 to 26]

8. Secondary Outcome: Hospital Free Days
Description: days alive and not admitted to a hospital;composite of hospital length of stay and death
Time Frame: from time of first eligibility to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
days | 2 [0 to 19] | 0 [0 to 17] | 0.5 [0 to 20] | 2 [0 to 19] | 0 [0 to 18]

9. Secondary Outcome: Ventilator Free Days
Description: days alive and not on mechanical ventilation; composite of ventilator free days and death
Time Frame: from time of first eligiblity to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
days | 22 [0 to 29] | 23 [0 to 29] | 21 [0 to 28] | 25 [1 to 29] | 21.5 [0 to 28]

10. Secondary Outcome: Hospital Discharge Disposition
Description: Location to which the patient was discharged after the end of the hospital admission
Time Frame: At the time of discharge from the hospital, up to 720 hours (30 days) after initiation of mechanical ventilation in a study ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
Participants
  ACH | 188 | 63 | 63 | 108 | 100
  EXPIRED | 844 | 264 | 231 | 367 | 394
  HOME | 954 | 310 | 228 | 488 | 354
  HOSPICE | 133 | 30 | 37 | 50 | 43
  OTHER | 26 | 8 | 9 | 5 | 12
  REHAB | 459 | 177 | 52 | 270 | 123
  SNF | 372 | 104 | 114 | 192 | 170

11. Secondary Outcome: Early Deep Sedation
Description: The percentage of time during the first 72 hours of mechanical ventilation that patients were alive, in the ICU, and with Richmond Agitation-Sedation Scale (RASS) of -3 to -5 . The RASS measures a patient's depth of sedation and ranges from -5 (comatose) to +4 (combative), with a normal level of 0 (defined as "alert and calm"). Negative values indicate a patient is sedated and positive values indicate some degree of agitation.
Time Frame: up to 72 hours, from the initiation to the discontinuation of mechanical ventilation in the ICU
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- Default Order Set + RT-targeted Accountable Justification: This arm will have the default order set and respiratory therapist-targeted accountable justification
  RT-targeted accountable justification: This strategy will require that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg into the flowsheet, similar to the physician-targeted accountable justification strategy.
  Default order set: With the default order set strategy, some mechanical ventilation order settings will be pre-populated to be consistent with LPV, including the mode and tidal volume, automatically calculated as 6 cc/kg of the patient's ideal body weight (as determined by each patient's height and gender, which are entered into the EHR on admission). The physician will have the option to opt out of any of the specified LPV settings and select other values.
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2953 | 949 | 725 | 1473 | 1189
percentage of time | 33 [3 to 93] | 33 [15 to 100] | 33 [0 to 83] | 33 [16 to 100] | 33 [0 to 91]

12. Secondary Outcome: Average Sedation Intensity Within the First 72 Hours
Description: Average Richmond Agitation-Sedation Scale (RASS) value, weighted by duration of time at that value. The RASS measures a patient's depth of sedation and ranges from -5 (comatose) to +4 (combative), with a normal level of 0 (defined as "alert and calm"). Negative values indicate a patient is sedated and positive values indicate some degree of agitation.
Time Frame: Up to 72 hours, from initiation to discontinuation of mechanical ventilation in a study ICU
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2953 | 949 | 725 | 1473 | 1189
score on a scale | -2.09 [-3.44 to -1.88] | -2.56 [-3.89 to -1.62] | -1.8 [-3.02 to -0.92] | -2.59 [-3.81 to -1.47] | -1.99 [-3.24 to -1.09]

13. Secondary Outcome: Deep Sedation for the Entirety of the First 72 Hours of Mechanical Ventilation
Description: Binary variable for whether a patient had Richmond Agitation-Sedation Scale (RASS) score of -3 to -5 for the entirety of the first 72 hours of mechanical ventilation. The RASS measures a patient's depth of sedation and ranges from -5 (comatose) to +4 (combative), with a normal level of 0 (defined as "alert and calm"). Negative values indicate a patient is sedated and positive values indicate some degree of agitation.
Time Frame: up to 72 hours, from initiation until discontinuation of mechanical ventilation in a study ICU
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
Number analyzed (Participants) | 2976 | 956 | 734 | 1480 | 1196
Participants
  Yes | 594 | 264 | 119 | 392 | 229
  No | 2362 | 687 | 609 | 1083 | 962
  Missing | 20 | 5 | 6 | 5 | 5

ADVERSE EVENTS:
Time Frame: All adverse events collected through 24 hours after study enrollment, which was defined as start of invasive mechanical ventilation in a study ICU. In addition, All-Cause Mortality was assessed through hospital discharge, up to 720 hours (i.e., 30 days), reported as outcome #6.
Description: Serious adverse events included (1) life threatening acidemia (pH <7.10), (2) mortality, or (3) cardiac arrest, all of which commonly occur in critically ill mechanically ventilated patients. Events were identified through daily reports reviewed by research coordinators and clinical experts to determine treatment-relatedness. Because this determination could be uncertain, we specified a priori that we would report all events in control and intervention groups for comparative purposes.
Groups:
- Physician-targeted Accountable Justification + RT-targeted Accountable Justification: This arm will have the physician-targeted accountable justification order set and respiratory therapist-targeted accountable justification flowsheet
  physician-targeted accountable justification: When a physician enters a mechanical ventilation order for a tidal volume that is greater than 6 cc/kg ideal body weight, an alert will appear requiring the physician to enter a reason for choosing a setting inconsistent with LPV. Clinicians will be instructed to provide a reason for deviation from LPV settings and that their response will be maintained in the medical record. The physician will not be able to sign the mechanical ventilation order set until after a response is entered.
  RT-targeted accountable justification: This strategy will require that the RT enter an explicit rationale in the EHR if he/she enters a tidal volume value greater than 6 cc/kg into the flowsheet, similar to the physician-targeted accountable justification strategy.
Arm/Group | Standard of Care | Default Order Set | Physician-targeted Accountable Justification | Default Order Set + RT-targeted Accountable Justification | Physician-targeted Accountable Justification + RT-targeted Accountable Justification
All-Cause Mortality (participants affected / at risk) | 844/2976 | 264/956 | 231/734 | 367/1480 | 394/1196
Serious Adverse Events (participants affected / at risk) | 95/2976 | 24/956 | 39/734 | 42/1480 | 64/1196
Other Adverse Events (participants affected / at risk) | 0/2976 | 0/956 | 0/734 | 0/1480 | 0/1196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=2976) | Default Order Set (N=956) | Physician-targeted Accountable Justification (N=734) | Default Order Set + RT-targeted Accountable Justification (N=1480) | Physician-targeted Accountable Justification + RT-targeted Accountable Justification (N=1196)
life-threatening acidemia (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 13 (13) | 18 (18) | 19 (19) | 27 (27) — pH less than 7.10 in the first blood gas after study enrollment, within 24 hours
mortality within 24 hours (Respiratory, thoracic and mediastinal disorders) | 50 (50) | 9 (9) | 19 (19) | 18 (18) | 29 (29) — All-cause mortality within 24 hours of study enrollment
cardiac arrest within 24 hours (Cardiac disorders) | 17 (17) | 2 (2) | 2 (2) | 5 (5) | 8 (8) — cardiac arrest, within 24 hours of study enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT04663802/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT04663802/SAP_001.pdf